CLINICAL TRIAL: NCT05206773
Title: A Randomized, Double-blind, Placebo-controlled, 12-month Phase 3 Study to Evaluate the Effect of Venglustat on Neuropathic and Abdominal Pain in Male and Female Participants ≥16 Years of Age With Fabry Disease Who Are Treatment-naïve or Untreated for at Least 6 Months
Brief Title: A Study to Evaluate the Effect of Venglustat Tablets on Neuropathic and Abdominal Pain in Male and Female Participants ≥16 Years of Age With Fabry Disease
Acronym: PERIDOT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC17045; U1111-1256-9310 (Registry Identifier: ICTRP); 2024-511990-31 (Registry Identifier: CTIS); 2021-002350-90 (EudraCT Number)
Record Dates: First submitted 2021-10-20; First posted 2022-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — venglustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants enrolled in the open-label extension will be treated with venglustat only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venglustat (Experimental): Participant will receive venglustat dose once daily for 12 months
  Interventions: Drug: Venglustat (GZ402671)
- Placebo (Placebo Comparator): Participants will receive placebo once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venglustat (GZ402671) — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Venglustat
Drug: Placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
This is a 12-month, parallel treatment, Phase 3, double-blind, randomized, placebo-controlled study to evaluate the effect of venglustat on neuropathic and abdominal pain symptoms of Fabry disease in participants ≥16 years of age with Fabry disease who are treatment-naïve or untreated for at least 6 months.

* Study visits will take place approximately every 3 months.
* The double-blind period will be followed by an open-label extension (OLE) during which participants who have completed the double-blind period will be treated with venglustat for an additional 12 months or until the Common Study End of Treatment Day (CSEOTD).

DETAILED DESCRIPTION:
Double blind period: the total duration will be up to approximately of 14 months (1 month of screening 12 month of treatment period, and a possible follow-up period of 1 month if no participation in the open label extension period)

Open-label extension period: the total duration will be approximately of 46 months (12 month of OLE treatment, additional OLE treatment until a common study end of treatment date (CSEOTD, approximately 33 months), and 1 month of follow-up period)

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients 16 year of age or older, who have had a previously confirmed diagnosis of Fabry disease and a history of clinical symptoms of Fabry disease
* Patients who are treatment-naïve or without prior treatment with an approved or experimental therapy for Fabry disease within at least 6 months prior to screening.
* Average score of ≥3 (0=no symptom, 10=symptom as bad as you can imagine) on the participant-defined most-bothersome symptom (among neuropathic pain in upper extremities, neuropathic pain in lower extremities, or abdominal pain), as measured by the Fabry Disease Patient-Reported Outcome (FD-PRO) at screening.
* Contraception (with double contraception methods) for male and female participants; not pregnant or breastfeeding for female participants; no sperm donation for male participants.
* Weight ≥30 Kg
* A signed informed consent must be provided prior to any study-related procedures.

Exclusion Criteria:

* Any manifestations of Fabry disease that preclude placebo administration.
* History of transient ischemic attack, stroke, myocardial infarction, heart failure, evidence of left ventricular hypertrophy and/or cardiac fibrosis, major cardiovascular surgery, or kidney transplantation.
* History of clinically significant cardiac arrhythmia. Atrial fibrillation that is well controlled on a stable medical regimen for at least 12 months is not an exclusion if the CHA2DS2-VASc score is 0 for males or 1 for females.
* Patients with hepatitis C, HIV, or hepatitis B infection.
* Neuropathic pain in upper or lower extremities, or abdominal pain not related to Fabry disease.
* History of seizures currently requiring treatment.
* Uncontrolled hypertension over the past 12 months prior to screening, or systolic BP >=150 or diastolic BP >=100 at screening.
* Estimated glomerular filtration rate <60 mL/min/1.73m².
* Urine protein to creatinine ratio >= 1 g/g at screening.
* Presence of severe depression as measured by Beck's Depression Inventory (BDI)-II >28 and/or a history of an untreated, unstable major affective disorder within 1 year of the screening visit.
* Positive SARS-CoV-2 virus test within 2 weeks of enrollment, or COVID 19 requiring hospitalization within 6 months of enrollment.
* Moderate to severe hepatic impairment.
* History of drug and/or alcohol abuse.
* History of or active hepatobiliary disease.
* Liver enzymes (alanine aminotransferase (ALT)/aspartate aminotransferase (AST)) or total bilirubin >2 times the upper limit of normal (ULN).
* Initiation of chronic treatment for pain, or change in pain medication regimen, within 3 months prior to randomization.
* Strong or moderate inducers or inhibitors of cytochrome P450 3A within 14 days or 5 half-lives, whichever is longer, prior to randomization.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline at 6 months in the most bothersome symptom of 3 Fabry Disease Patient-Reported Outcome (FD-PRO) items (neuropathic pain in upper extremities, neuropathic pain in lower extremities, or abdominal pain) | From baseline to 6 months
Percent change from baseline at 12 months in the most bothersome symptom of 3 Fabry Disease Patient-Reported Outcome (FD-PRO) items (neuropathic pain in upper extremities, neuropathic pain in lower extremities, or abdominal pain) | From baseline to 12 months

SECONDARY OUTCOMES:
Percent change in plasma globotriaosylsphingosine (lyso-GL-3) | From baseline to 6 month and 12 months
Frequency of rescue pain medication use | From baseline to 6 months and 12 months
  Number of days with use of rescue pain medications during the 6-month treatment period, divided by duration of the 6-month treatment period and multiplied by 100. The same definition will be used for the 12-month period.
Change in the percentage of days with at least 1 stool reflecting diarrhea (Bristol Stool Form Scale [BSFS] Type 6 or 7) | From baseline to 6 month and 12 months
Change in tiredness component of FD-PRO | From baseline to 6 month and 12 months
Proportion of responders in neuropathic or abdominal pain, as assessed by FD-PRO | At 6 months and 12 months
  Response is defined as at least a 30% decrease from baseline in the most bothersome of 3 FD-PRO items between neuropathic pain in upper extremities, neuropathic pain in lower extremities, and abdominal pain
Number of participants with adverse event (AE) and serious adverse event (SAE) | From baseline to 6 month and 12 months
Change in the lens clarity (new or worsening lens opacities) by ophthalmological examination (by slit lamp exam at Visit 2 and Visit 6) | From baseline to 12 months
Change in Beck Depression Inventory-II (BDI-II) score | From baseline to 6 month and 12 months
Plasma venglustat concentrations at prespecified visits over the study duration | From baseline to 6 month and 12 months
Maximum venglustat plasma concentration (Cmax) | From baseline to 6 month and 12 months
Time to maximum venglustat plasma concentration (tmax) | From baseline to 6 month and 12 months
Area under the venglustat plasma concentration versus time curve from time 0 to 24 hours (AUC0-24) | From baseline to 6 month and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (58):
- United States (12):
  - Nephrology Clinic at Kirklin Clinic of UAB Hospital_Investigational Site Number: 8400011, Birmingham, Alabama
  - UCLA Medical Center_Investigational Site Number: 8400006, Los Angeles, California
  - University of California Irvine Medical Center- Site Number : 8400019, Orange, California
  - Advent Health Orlando_Investigational Site Number: 8400008, Orlando, Florida
  - Emory Genetics- Site Number : 8400010, Atlanta, Georgia
  - Westchester Medical Center Healthcare Corporation- Site Number : 8400001, Hawthorne, New York
  - Cincinnati Children's Hospital Medical Center - PIN- Site Number : 8400013, Cincinnati, Ohio
  - Cleveland Clinic Site Number : 8400016, Cleveland, Ohio
  - Children's Hospital Of Pittsburgh- Site Number : 8400009, Pittsburgh, Pennsylvania
  - Renal Disease Research Institute, An affiliate of: Dallas Nephrology Associates_Investigational Site Number: 8400012, Dallas, Texas
  - University Of Utah Health Sciences Center- Site Number : 8400005, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center_Investigational Site Number: 8400004, Fairfax, Virginia
- Argentina (2):
  - Fundacion Cori para la Investigación y Prevención del Cancer_Investigational Site Number: 0320002, La Rioja
  - Instituto de Investigaciones Clínicas Quilmes (IICQ) SRL_Investigational Site Number: 0320003, Quilmes
- Investigational Site Number : 0360001, Parkville, Victoria, Australia
- Investigational Site Number: 0400001, Vienna, Austria
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre_Investigational Site Number: 0760001, Porto Alegre, Rio Grande do Sul
  - Instituto de Genética e Erros Inatos do Metabolismo - IGEIM- Site Number : 0760002, São Paulo
- Canada (3):
  - M.A.G.I.C Calgary LTD_Investigational Site Number: 1240003, Calgary, Alberta
  - Medicine Dalhousie University_Investigational Site Number : 1240001, Halifax, Nova Scotia
  - University Health Network_Investigational Site Number : 1240005, Toronto, Ontario
- China (4):
  - No.8, Xishiku Street, Xicheng District_Site Number: 1560001, Beijing
  - No.197,2nd Ruijin road, Huangpu district_Site Number: 1560003, Shanghai
  - No.85 South Jiefang road, Yingze District_Site Number: 1560004, Taiyuan
  - Investigational Site Number : 1560006, Zhengzhou
- Investigational Site Number: 2080001, Copenhagen, Denmark
- Investigational Site Number: 2460001, Turku, Finland
- Investigational Site Number : 2500001, Garches, France
- Germany (4):
  - ISphinCS GmbH_Investigational Site Number: 2760004, Hochheim am Main
  - Investigational Site Number : 2760005, Mainz
  - Investigational Site Number: 2760003, München
  - Investigational Site Number: 2760001, Würzburg
- Greece (3):
  - Investigational Site Number : 3000003, Athens
  - University Hospital of Heraklion_Investigational Site Number: 3000001, Heraklion
  - University Hospital of Ioannina_Investigational Site Number: 3000002, Ioannina
- Italy (5):
  - IRCCS Policlinico di Sant'Orsola_Investigational Site Number : 3800005, Bologna
  - Fondazione IRCCS San Gerardo dei Tintori, S.C. Nefrologia - Clinica Nefrologica_Investigational Site Number: 3800002, Monza
  - Azienda Ospedaliera Universitaria "Federico II", U.O. di Nefrologia- Diparimento di Sanità Pubblica_Investigational Site Number: 3800001, Napoli
  - Azienda Ospedaliera Universitaria_Investigational Site Number: 3800003, Palermo
  - Fondazione Policlinico Universitario_Investigational Site Number: 3800004, Roma
- Japan (4):
  - Investigational Site Number : 3920005, Kawasaki, Kanagawa
  - Fukuoka University Hospital_Investigational Site Number: 3920004, Fukuoka-shi, Fukuoka
  - The Jikei University Hospital_Investigational Site Number: 3920003, Minato-ku, Tokyo
  - Tohoku University Hospital_Investigational Site Number: 3920001, Sendai-shi, Miyagi
- Mexico (2):
  - Hospital Universitario "Dr. José Eleuterio González" Departamento de Genética Centro Universitario contra el cáncer_Investigational Site Number: 4840001, Monterrey, Nuevo León
  - Odette del Carmen DIAZ-AVENDAÑO Clinstile, S.A. de C.V. Durango_Investigational Site Number: 4840002, Mexico City
- Investigational Site Number: 5780001, Bergen, Norway
- Poland (3):
  - Investigational Site Number : 6160002, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160004, Rzeszów
  - Investigational Site Number: 6160003, Wroclaw
- Institutul Clinic Fundeni_Investigational Site Number: 6420001, Bucharest, Romania
- Investigational Site Number : 7560001, Zurich, Switzerland
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920002, İzmit
  - Investigational Site Number : 7920004, Malatya
- United Kingdom (3):
  - Investigational Site Number: 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number: 8260002, London, London, City of
  - Investigational Site Number : 8260003, Salford, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17045 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25261&tenant=MT_SNY_9011